CLINICAL TRIAL: NCT03735602
Title: The Research of the Neural Mechanisms Underlying Astigmatism
Brief Title: Neural Mechanisms Underlying Astigmatism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Clinical Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JYuan
Record Dates: First submitted 2018-10-24; First posted 2018-11-08 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- perceptual training (Experimental): Orientation discrimination task, which is a cognitive task. Patients were trained for 1 hour per day, 15 days in total.
  Interventions: Behavioral: perceptual training

INTERVENTIONS:
Behavioral: perceptual training — orientation discrimination task

SUMMARY:
This study is to compare the contrast sensitivity function and neural response to gratings before and after the orientation discrimination task in the astigmatism or amblyopia patients.

DETAILED DESCRIPTION:
The presence of astigmatism can lead to substantial reductions in visual performance in a variety of clinical vision measures and functional visual tasks. However, the neural mechanisms underlying the astigmatism remains unknown. The current study recruited three groups (patients with with-the-rule astigmatism and amblyopia, patients with with-the-rule astigmatism but without amblyopia, normal controls) of subjects and patients receive perceptual learning training (orientation discrimination task) which lasts for around 15 days. This main aim is to compare the contrast sensitivity function and neural response to gratings before and after the orientation discrimination task in the astigmatism or amblyopia patients.

Patients with astigmatism or amblyopia were included in this study. All participants underwent an ophthalmic examination that included slit-lamp biomicroscopy, visual acuity, quick CSF under full optical correction, 9-SF life quality questionnaire and fundus examination.

ELIGIBILITY:
Inclusion Criteria:

* high astigmatism

Exclusion Criteria:

* other types of disease (especially optical diseases) that may affect study

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The change of the contrast sensitivity function tested by quick CSF | eight months
  The quick CSF (contrast sensitivity function) measures contrast threshold by fitting raw data and calculating the Cutoff sensitivity frequency.
The change of contrast threshold tested by sweep visually evoked potential (VEP) | eight months
  The contrast threshold was calculated by analyzing EEG(Electroencephalogram) data recorded with sweep visually evoked potential (VEP) paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yuan, Professor, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided